CLINICAL TRIAL: NCT00269425
Title: The Heart Institute of Spokane Diet Intervention and Evaluation Trial (THIS DIET)
Brief Title: The Heart Institute of Spokane Diet Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: The Heart Institute of Spokane (Unknown); Providence Medical Research Center (Other); Washington State Attorney General's Office (Other); Deaconess Medical Center, Spokane, Washington (Other)
Responsible Party: Katherine R. Tuttle, MD, Providence Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THIS-A20010724157261
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2005-12

CONDITIONS: Myocardial Infarction
Keywords: Cardiovascular disease; Nutrition; Mediterranean diet; Low fat diet; American Heart Association diet; Monounsaturated fats; Omega-3 fats; Outcomes
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases | interventions — Diet, Fat-Restricted; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mediterranean diet, (Experimental)
  Interventions: Behavioral: Mediterranean diet
- American Heart Association Step 2 diet (Experimental)
  Interventions: Behavioral: American Heart Association Step 2 diet
- Case controlled (No Intervention)

INTERVENTIONS:
Behavioral: American Heart Association Step 2 diet — Low fat diet with patient education and diet analysis
  Other Names: Low fat diet
  Arms: American Heart Association Step 2 diet
Behavioral: Mediterranean diet — Mediterranean style diet with patient education and diet analysis
  Arms: Mediterranean diet,

SUMMARY:
The purpose of this study is to determine whether a Mediterranean style diet, enriched in monounsaturated and omega-3 fats, is superior to the American Heart Association Step 2 diet, a traditional low fat diet, for improving rates of survival and cardiovascular complications in persons who have had a first myocardial infarction (heart attack).

DETAILED DESCRIPTION:
Cardiovascular diseases (heart attack, stroke, and other vascular diseases) are major causes of mortality in developed countries. Although medicines and revascularization procedures prolong lives, rates of death and disability remain high. Lifestyle factors greatly contribute to risk. Yet, scientific data regarding the role of lifestyle change in prevention and treatment are limited. In the nutrition area, limitations include observational or uncontrolled study design, and focus on surrogate markers rather than on clinical outcomes.

Excess dietary fat has long been associated with cardiovascular diseases. Increased risk is related both to types of fat and calories from fat. Saturated fat, cholesterol, and trans-fatty acids have all been associated with adverse outcomes. Because fat is calorie-laden, high fat diets are commonly associated with weight gain and obesity. Low-fat diets have traditionally been recommended to control lipids and weight. However, these diets are high in carbohydrate and may actually be associated with weight gain if calories are not limited. Such diets have also been associated with worsening of hyperinsulinemia and insulin resistance and an adverse lipid pattern (low HDL cholesterol and high triglyceride levels). In contrast, increased intake of monounsaturated and omega-3 fats is associated with favorable effects on cardiovascular risk factors and markers including: endothelial function, lipids, and levels of insulin and glucose. Results have been consistent across various groups of high-risk patients, including those with hypercholesterolemia, diabetes, and hypertension. Most importantly, a Mediterranean style diet enriched in monounsaturated and omega-3 fats reduced death and cardiovascular complications after myocardial infarction (MI) in the Lyon Heart study.

The American Heart Association (AHA) Step 2 is a low-fat diet traditionally recommended for people with cardiovascular disease. The Mediterranean and AHA Step 2 diets differ primarily in the amount of monounsaturated and omega-3 fats, both of which are higher in the Mediterranean diet. Both diets are low in saturated fat (less than 7%) and cholesterol (less than 200 mg/d). Although the Lyon Heart Study compared a Mediterranean diet to a "prudent Western diet," a low fat diet similar to the AHA diet, the latter group did not achieve recommended intake levels of saturated fat or cholesterol. Furthermore, there was no longitudinal nutritional intervention in the low fat diet group. Therefore, the effect of nutritional intervention per se was not addressed.

Comparison(s): In survivors of a first MI, two longitudinal nutritional interventions, a Mediterranean style diet and an AHA Step 2 diet, will be compared. Both intervention groups will be compared to an untreated control group from our clinical database.

ELIGIBILITY:
Inclusion Criteria:

* First myocardial infarction

Exclusion Criteria:

* Prior myocardial infarction
* Uncontrolled or secondary hypertension
* New York Heart Association heart failure stage III or IV
* Ventricular arrythmias requiring medical or defibrillatory intervention
* Other diseases that may make study completion difficult or unlikely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2000-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Fatal/non-fatal myocardial infarction | 3,6,12,18,24,36,48,60,72 months
  The primary outcome was a composite of end points including all-cause and cardiac deaths, MI, hospital admissions for heart failure, unstable angina, or stroke.
Cardiovascular death | 3,6,12,18,24,36,48,60,72 months
Non-cardiovascular death | 3,6,12,18,24,36,48,60,72 months
Stroke/TIA | 3,6,12,18,24,36,48,60,72 months
Admission for congestive heart failure or unstable angina | 3,6,12,18,24,36,48,60,72 months

SECONDARY OUTCOMES:
Cardiovascular revascularization | 3,6,12,18,24,36,48,60,72 months
Peripheral revascularization or amputation | 3,6,12,18,24,36,48,60,72 months
Doubling of serum creatinine,dialysis,or kidney transplant | 3,6,12,18,24,36,48,60,72 months
New hypertension | 3,6,12,18,24,36,48,60,72 months
New diabetes | 3,6,12,18,24,36,48,60,72 months
Risk factors (traditional and novel) | 3,6,12,18,24,36,48,60,72 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine R. Tuttle, MD,FASN,FACP, Principal Investigator — Providence Medical Research Center
Locations (1):
- Providence Medical Research Center, Spokane, Washington, United States